CLINICAL TRIAL: NCT05353855
Title: Neural Correlates of Impulsivity in Idiopathic REM Sleep Behavior Disorder: a Functional Magnetic Resonance Imaging Case-control Study
Brief Title: Neural Correlates of Impulsivity in Idiopathic REM Sleep Behavior Disorder
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: HMRF08191416
Record Dates: First submitted 2022-01-13; First posted 2022-04-29 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Impulsivity; Prodromal Parkinson's disease; REM sleep behavior disorder; Functional Magnetic Resonance Image
MeSH Terms: conditions — Parkinson Disease; Impulsive Behavior; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early unmedicated PD patients converted from iRBD: 1. Chinese aged 50 or above;
  2. Being capable of giving informed consent for participation of the study;
  3. Having a diagnosis of PD confirmed by neurologists according to the United Kingdom Parkinson's Disease Survey Brain Bank.
  4. Onset of PD motor symptoms of < 3 years;
  5. In view of the heterogeneity of PD, the investigator will only include those patients with RBD preceding the onset of motor symptoms of PD.
  6. Drug naïve (dopaminergic medications have not been started)
  Interventions: Other: No intervention
- Early medicated PD patients converted from iRBD: Inclusion criteria will be the same as that of early unmedicated PD except that they should be on dopaminergic medications.
  Interventions: Other: No intervention
- iRBD patients: 1. Chinese aged 50 or above;
  2. Being capable of giving informed consent for participation of the study;
  3. Having a diagnosis of RBD according to the International classification of sleep disorder 3rd edition (ICSD 3rd), fulfilling both the clinical and video-polysomnography (vPSG) criteria.
  Interventions: Other: No intervention
- Healthy controls: 1. Age-and sex-matched with the groups;
  2. Being capable of giving informed consent for participation of the study;
  3. Without a personal history or a family history of PD or RBD;
  4. A total score on REM Sleep Behavior Questionnaire (RBDQ-HK) less than 19, which is the suggestive cut-off of a diagnosis of RBD;
  5. Absence of self-report dream enactment behaviors and RSWA as measured by v-PSG.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aims to investigate the neural correlates (structural changes, functional connectivity, and structural connectivity of brain structures in prefrontal cortex and basal ganglia) of impulsivity by measuring structures and the blood-oxygen-level-dependent signal of brain in response to impulsive tasks and task-free using functional Magnetic Resonance Image method among healthy controls, patient with prodromal PD (iRBD), and patients with PD.

DETAILED DESCRIPTION:
Background: Excessive impulsivity is an important non-motor symptom of Parkinson's disease (PD), especially for those on dopamine agonist treatment. Dopaminergic dysfunction has been highly correlated with impulsivity. Given that idiopathic REM sleep behavior disorder (iRBD) is a prodromal stage of alpha-synucleinopathy, such as PD, the dysfunction of dopaminergic system at this early stage may also precipitate alternation of impulsivity.

Hypothesis and objectives: iRBD may have altered impulsivity which is similar to that found in de novo PD and may serve as a biomarker in differentiating iRBD from healthy controls. This study aims to investigate the neural correlates (structural changes, functional connectivity, and structural connectivity of brain structures in prefrontal cortex and basal ganglia) of impulsivity by measuring structures and the blood-oxygen-level-dependent signal of brain in response to impulsive tasks and task-free using functional Magnetic Resonance Image method among healthy controls, patient with prodromal PD (iRBD), and patients with PD.

Design and subjects: This is a case-control study that will recruit 96 subjects (24 healthy controls, 24 patients with iRBD, 24 PD patients on dopaminergic medication and 24 PD patients who are not on dopaminergic medication).

Main outcome measures: 1) The difference in brain activity in response to impulsivity tasks between groups; 2) The difference in structure volume, structural and functional connectivity of region of interest related to impulsivity (prefrontal cortex and basal ganglia) between groups; 3) The association of these changes with the stage of disease from healthy, to prodromal, and to clinically diagnosed PD.

ELIGIBILITY:
Inclusion Criteria:

1. Age-and sex-matched with the groups;
2. Being capable of giving informed consent for participation of the study;
3. Without a personal history or a family history of PD or RBD;
4. A total score on REM Sleep Behavior Questionnaire (RBDQ-HK) less than 19, which is the suggestive cut-off of a diagnosis of RBD;
5. Absence of self-report dream enactment behaviors and RSWA as measured by v-PSG

Exclusion Criteria:

1. Having a history of ICD diagnosis or ICD symptom(s) assessed with Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS);
2. Presence of narcolepsy or other neurodegenerative diseases (except for PD group) that may give rise to RBD;
3. Presence of mood disorder which may have great impact on impulsivity;
4. A total score of the Montreal Cognitive Assessment (MOCA) ≤ 22 and the Clinical Dementia Rating (CDR) ≥ 1, indicating dementia;
5. Except for early medicated PD patients, if subjects from other groups who are on medication that may induce impulsivity, such as dopaminergic medication, will be excluded;
6. Contraindication to MRI (e.g., presence of implants or claustrophobia).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a case-control study. We plan to recruit four groups of participants: patients with PD on/are not on dopaminergic medication converted from iRBD, patients with iRBD, and healthy control group.
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain activity | 1 year
  To access different cognitive aspects in neurobehavioral impulsivity such as BART, TCIP and SKIP between groups

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Data will be handled and stored under Department of Psychiatry and PI will be responsible for the safekeeping.